CLINICAL TRIAL: NCT00706875
Title: A Global Assessment of Medical, Emotional and Reproductive Concerns in Gestational Trophoblastic Disease Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-040
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Uterine Cancer; Cervix Uteri Nos; Gestational Trophoblastic Disease
Keywords: GTD survivors; questionnaires; GTD
MeSH Terms: conditions — Uterine Neoplasms; Gestational Trophoblastic Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 1: 30 patients survived GTD post treatment for 0 - 5 years.
  Interventions: Behavioral: questionnaire
- 2: 30 patients survived GTD post treatment 6 - 10+ years.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — A patient questionnaire, which includes validated instruments. Data collection methods are as follows:
  * In person at the medical appointment
  * Over the telephone
  * Mailed with self-addressed return envelope and prepaid postage
  * E-mailed and returned by e-mail, fax or self-addressed envelope and pre-paid postage
  Groups: 1
Behavioral: questionnaire — A patient questionnaire, which includes validated instruments. Data collection methods are as follows:
  * In person at the medical appointment
  * Over the telephone
  * Mailed with self-addressed return envelope and prepaid postage
  * E-mailed and returned by e-mail, fax or self-addressed envelope and pre-paid postage
  Groups: 2

SUMMARY:
The purpose of this study is to collect information on the effects of treatment for gestational trophoblastic disease (GTD). We plan to use the findings from this study to better understand GTD survivors' health and quality of life.

We would like to know more about the health, quality of life and pregnancies of women treated for GTD. This information will be used to try and improve the treatments for women who have this disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed GTD by MSKCC
* Sufficient proficiency in the English language to respond to quality of life surveys
* Age ≥ 18 years
* Benign or malignant disease
* Treated with surgery and/or chemotherapy or observation

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: GTD survivors treated at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The primary outcomes include reproductive concerns (as measured by the Reproductive Concern Scale, RCS) and sexual functioning (as measured by the Female Sexual Function Index, FSFI). | conclusion of the study

SECONDARY OUTCOMES:
To describe the prevalence of premature menopause and increased bone loss through the Menopausal Symptom Check List and medical follow-up information. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jewell, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org